CLINICAL TRIAL: NCT07303569
Title: Prevention of Pressure Injury (PI) in Hospitalised Infants, Children, and Young People (CYP) (Aged 0-19 Years)
Acronym: CYPPI
Status: Recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Leicester (Other); University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: 24CS003
Record Dates: First submitted 2025-09-19; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Pressure Injuries; Pressure Ulcers, Bedsores, Decubitus Ulcer
Keywords: Pressure Injury prevention; assessment; tools (instruments); Validity; Dark skin tone
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
What is the problem? Children and young people admitted to hospital can sometimes be harmed by what is called a pressure injury. Pressure injuries are sores (ulcers) that happen on areas of the skin that are under pressure. The pressure can come from lying in bed, sitting in a wheelchair, or wearing a cast for a long time. They usually form on bony parts of the body, such as the heels, elbows, hips, and tailbone. This can be uncomfortable for the patient and distressing for their families. As well, it means that more staff and treatments are needed for the patient.

What is known? There is a difference in pressure injury seriousness for infants and children with dark skin tones to those without. Pressure injury care for hospitalised patients starts with an assessment using a tool. In the past, the assessment tools were developed without consideration for differences due to skin tone. This means that the current tools may not be the best way to identify pressure injury for dark skin tones. Healthcare professionals need to make sure that tools are fit for purpose for all.

What are investigators going to do? Investigators will work with healthcare professionals, children, and parents together to develop and test the existing pressure injury risk assessment tool for use with dark skin tones.

This study is a result of care priority discussions with parents and children. It came from the patients and will benefit the patients. Children, young people, and parents will be involved throughout to ensure their voices are heard.

How are investigators going to do it?

Investigators will:

1. Look at existing information about pressure injury for children with darker skin tones. If required, investigators will change and increase the accuracy of the existing tool.
2. Test the modified risk assessment tool at 10 children's hospitals in the UK. Investigators will do this to see if it can distinguish hospitalised children with dark skin tones, at high or low risk of pressure injury development during their hospital stay.

DETAILED DESCRIPTION:
Research Question/Aim(s): How accurate is the BRADEN-QD in capturing risk of pressure injury (PI) in hospitalised infants and children and young people (CYP) with dark skin tones (DST)? Aim: To evaluate critical gaps in knowledge and evidence by modification (as required) and validation of the BRADEN-QD in hospitalised infants and CYP with DST.

Objectives:

1. To identify and gain consensus on additional factors pertinent to hospitalised CYP with DST for inclusion in the BRADEN-QD [Phase 1].
2. To validate the original/modified BRADEN-QD in a DST population through multi-centre study [Phase 2].

Study Design This is a mixed methods sequential study comprising of two phases; Phase 1 (information gathering) consists of two Work Packages (WPs 1 and 2). WP1: Individual interviews or focus groups with stakeholders to identify further PI risk items not captured from the literature. Interviews will be conducted online, over the telephone or face-to-face according to participant preference. Interviews will be audio recorded and transcribed verbatim.

WP2: Participants from stage 1 are invited to take part in a 60-minute Nominal Group Technique online workshop to rank, according to relevance and importance, the PI risk items identified from stage 1. A modified Delphi technique will be used and items with a consensus of ≥ 70% will be added to the BRADEN-QD to create a modified BRADEN-QD (mBRADEN-QD).

Study Phase 2; A multicentre pyschometric validation approach will be used to assess the accuracy and validity of the original tool (BRADEN-QD) or modified BRADEN-QD tool (mBRADEN-QD), based on Phase 1 findings.

Study Participants Phase 1: WP1 and WP2: Healthcare professionals (HCP), Children and young people (CYP), and parents/ guardians.

Phase 2: Hospitalised CYP with dark skin tone. Planned Size of Sample (if applicable) Phase 1: WP1 total participants 20 (7 CYP, 7 parents/ guardians and 6 HCP). WP2 participants from WP1 will be invited to take part. A minimum of 10 participants required.

Phase 2: A total of 522 participants will be recruited into the study across 10 sites. Each site will be expected to recruit a total of 52 participants.

Follow up duration (if applicable): Phase 2 For participants recruited for Phase 2, PI assessment is to be completed three times per week (Monday, Wednesday and Friday) for two full weeks and then once weekly for two weeks = maximum 8 times total follow up. Subject data will be considered complete at discharge or hospital day 28 after enrolment into the study whichever occur first. Any identified hospital acquired pressure injuries (HAPIs) will be categorised according to stage and causation. HAPIs will be managed at the discretion of the clinical team.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

HCP participants:

1. Experts (e.g. tissue viability practitioners, dermatologist)
2. HCP looking after hospitalised infants and CYP
3. Able to give consent

Parent/ guardian participants:

1. Parents/ guardians of infants and CYP admitted to hospital with or developed PI
2. Parent/ guardian of a CYP under 19 years of age with dark skin tone according to Fitzpatrick Classification of Skin Types III, IV, V or VI.
3. Able to give consent

CYP participants:

1. Age 10 - 19
2. Dark skin tone according to Fitzpatrick Classification of Skin Types III, IV, V or VI.
3. Able to gain consent
4. Able to provide assent with parental consent
5. Developed PI during hospitalisation Phase 2 Hospitalised infants and CYP participants

1. Infants and CYP admitted to hospital for 24 hrs 2. Age 0-19 years 3. Able to gain consent. 4. Fitzpatrick Classification of Skin Types IV, V or VI.

Exclusion Criteria:

Phase1:

HCP participants:

1. HCP not working with hospitalised infants and CYP.
2. Unable to provide consent.

Parents participants:

1. Parents of hospitalised infants and CYP with no PI.
2. Unable to gain consent

CYP participants:

1. Not able to provide consent
2. CYP with no PI during hospitalisation period Phase 2

1. Admitted to hospital for less than 24 hrs 2. Unable to gain consent 3. Fitzpatrick Classification of Skin Types I, II or III

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Phase 1: Healthcare professionals who look after infants, children and young people in hospital (children's nurses and doctors from various clinical areas, dermatologist, tissue viability practitioners and clinical educators); parents/ guardians of children who have a dark skin tone, have developed a pressure injury(s) while in hospital before, and children and young people with dark skin tones who have developed pressure injury(s) while in hospital before.
  Phase 2: Children and young people with dark skin tone admitted to hospital.
Sampling Method: Non-Probability Sample
Enrollment: 542 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-05-16 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Total PI risk assessment score measured using the BRADEN-QD scale with or without additional items | up to 4 weeks
  Total PI risk assessment score. The scale uses a 0 to 20 point scale, with scores of 13 or higher indicating a patient is at risk for a PI
Pressure Injury development | up to 4 weeks
  Developing a pressure injury while in hospital.

SECONDARY OUTCOMES:
Length of hospital stay (LOS) | up to 24 weeks
  Number of days in hospital
Morbidity | Up to 4 weeks
  Complications experienced while in hospital
Mortality | up to 4 weeks
  Deaths while in hospital
Economic impact | Up to 4 weeks
  Estimated treatment costs from pressure injury

CONTACTS AND LOCATIONS:
Overall Officials: Takawira C Marufu, Phd, Principal Investigator — Nottingham University Hospital
Locations (1):
- Nottingham University Hospital, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided